CLINICAL TRIAL: NCT07403110
Title: Effects of Kaltenborn Mobilization With and Without Proprioceptive Neuromuscular Facilitation Technique on Pain, Range of Motion and Function in Patients With Chronic Non Specific Low Back Pain.
Brief Title: Kaltenborn Mobilization With and Without Proprioceptive Neuromuscular Facilitation Technique in Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0177
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: disability; mobility; back pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaltenborn Mobilization with Proprioceptive neuromuscular facilitation technique (Experimental)
  Interventions: Other: Kaltenborn mobilization; Other: Proprioceptive Neuromuscular Facilitation Technique; Other: Standard Physiotherapy Treatment
- Kaltenborn mobilization (Active Comparator)
  Interventions: Other: Kaltenborn mobilization; Other: Standard Physiotherapy Treatment

INTERVENTIONS:
Other: Kaltenborn mobilization — Kaltenborn mobilization was applied to the lumbar spine area in the dorsal direction . Patient was positioned in flexion , side bending and rotation to the right and glide was applied in dorsal direction. Similar glide was given to patient in extension, side bending and rotation to the right. These techniques were performed for 3 days per week for 6 consecutive weeks.
Other: Proprioceptive Neuromuscular Facilitation Technique — PNF Hold Relax technique was performed on lumbar spine to increase the extensibility of the surrounding muscles after a maximal response. These techniques were performed for 3 days per week for 6 consecutive weeks.
  Arms: Kaltenborn Mobilization with Proprioceptive neuromuscular facilitation technique
Other: Standard Physiotherapy Treatment — Hotpack for 10 mins was applied with Tens at a burst mode with pulse width 200 microsec, frequency 100 Hz, burst frequency 2 Hz for 10 mins. Ultrasound was applied for 10 mins, stretching of calf, hamstrings and gluteals along with back strengthening.

SUMMARY:
The study was conducted to determine the effects of Kaltenborn mobilization with and without proprioceptive neuromuscular facilitation technique on pain, range of motion and function in patients with chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 25 to 45
* Pain lasting for more than 3 months
* Score between 2 to 7 in NPRS
* Score of greater than 20 in ODI
* Pain localized between the level below the ribs at the posterior side and above the level of buttocks.

Exclusion Criteria:

* Any neoplasm involving back
* Radiating pain
* Metabolic disorders like osteoporosis
* Pregnancy
* Acute infection
* Prior orthopedic surgeries
* Acute trauma

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-10-14 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | From enrollment to the end of treatment at 6 weeks.
  Numeric Pain Rating scale is used to measure intensity of pain. It ranges from 0 to 10 where 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain and 7-10 shows severe pain.
Oswestry Disability Index | From enrollment to the end of treatment at 6 weeks
  Oswetry Disability index is a questionnaire consisting of 10 questions used to asses functional disability in patients with low back pain. In this scale, 0-20% = minimal disability, 21-40% = moderate disability, 41-60% = severe disability, 61-80% = crippled and 81-100% = bedbound.

SECONDARY OUTCOMES:
ROM Lumbar spine (Flexion) | From enrollment to end of treatment at 6 weeks.
  Changes in lumbar flexion range of motion was measured using goniometer at baseline and at the end of 6 weeks.
ROM of Lumbar Spine ( Extension) | From enrollment to the end of treatment at 6 weeks
  Changes in lumbar extension range of motion was measured using goniometer at baseline to the end of treatment at 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Shakil ur Rehman, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- General Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panjaitan LA, Hon WHC, Baait SN, Mawaddah N. Comparison between proprioceptive neuromuscular facilitation and mckenzie method in lumbar range of motion on non-specific low back pain. ACTIVE: Journal of Physical Education, Sport, Health and Recreation. 2020;9(1):63-71.
- [Background] Mehyar F, Santos M, Wilson SE, Staggs VS, Sharma NK. Effect of grade III lumbar mobilization on back muscles in chronic low back pain: a randomized controlled trial. Journal of Allied Health. 2020;49(1):20-8.
- [Background] Thomas JS, Clark BC, Russ DW, France CR, Ploutz-Snyder R, Corcos DM; RELIEF Study Investigators. Effect of Spinal Manipulative and Mobilization Therapies in Young Adults With Mild to Moderate Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2012589. doi: 10.1001/jamanetworkopen.2020.12589. PMID 32756930
- [Background] Karkamandi F, Miri H, Letafatkar A, Haghighi M. Comparing the effects of motor control exercises and PNF exercises on postural control, strength, endurance, and proprioception in women with chronic nonspecific low back pain. Sport Sciences and Health Research. 2021;13(2):165-77.
- [Background] Fouda KZ, Dewir IM, Abdelsalam MS. Effects of proprioceptive neuromuscular facilitation techniques in treating chronic nonspecific low back pain patients. Physiotherapy Quarterly. 2021;29(2):32-7.
- [Background] Lizis P, Kobza W, Jaszczur-Nowicki J, Wisniewski D. Osteopathic Manual Treatment Compared to Kaltenborn-Evjenth Orthopedic Manual Therapy for Chronic Low Back Pain: A Randomized Study. Alternative Therapies in Health and Medicine. 2021:AT6593-AT.
- [Background] Koutarapu S, Ghumare D. Proprioceptive neuromuscular facilitation exercises versus lumbar stabilization exercises for chronic low back pain patients: A randomized interventional study. The Indian Journal of Occupational Therapy. 2022;54(1):23-8.
- [Background] Arcanjo FL, Martins JVP, Mote P, Leporace G, de Oliveira DA, de Sousa CS, et al. Proprioceptive neuromuscular facilitation training reduces pain and disability in individuals with chronic low back pain: A systematic review and meta-analysis. Complementary Therapies in Clinical Practice. 2022;46:101505.
- [Background] Malik A, Ramsha M, Samad A. Outcomes of the butler neural mo-bilization technique and manual therapy for chronic low back pain in patients with lumbar radiculopathy: A cross-sectional comparative study. J Basic Clin Med Sci. 2022;1:3-11.
- [Background] Kasimis K, Iakovidis P, Lytras D, Koutras G, Chatziprodromidou IP, Fetlis A, et al. Short-term effects of manual therapy plus capacitive and resistive electric transfer therapy in individuals with chronic non-specific low back pain: a randomized clinical trial study. Medicina. 2023;59(7):1275.
- [Background] Shahzadi M, Tanveer S, Batool M, Sheikh SA, Faraz K, Fatima Z. Comparing Muscle Energy Technique and Kaltenborn-Evjenth Orthopaedic Manual Therapy: A Study on Effectiveness in Treating Chronic Low Back Pain. Journal of Health and Rehabilitation Research. 2023;3(2):1200-5.
- [Background] Khalid R, Hasan S, Anis T, Riaz SW, Maroof A, Arshad A, et al. Comparative Effectiveness of Muscle Energy Technique (MET) With or Without Proprioceptive Neuromuscular Facilitation (PNF) Pattern in Lumbosacral Dysfunction: Comparative Effectiveness of Muscle Energy Technique (MET). THE THERAPIST (Journal of Therapies & Rehabilitation Sciences). 2024:51-5.
- [Background] Deopa V, Kumar N, Thapliyal S, Sharma S. To Compare the Effect of PNF Stretching and Core Stabilizing Exercise Versus McKenzie Technique in Subjects with Low Back Pain.